CLINICAL TRIAL: NCT02669979
Title: Domiciliary Professional Oral Care for Dependent Elderly - Access to Improved Oral and General Health?
Brief Title: Domiciliary Professional Oral Care for Dependent Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Inger Wårdh, PhD Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KarolinskaACT
Record Dates: First submitted 2016-01-19; First posted 2016-02-01 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Dental Caries; Gingivitis
Keywords: elderly; oral care
MeSH Terms: conditions — Dental Caries; Gingivitis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention in the research groups is professional oral care with tooth brush, "ordinary" fluoridated tooth paste (1100-1450 ppm NaF), and repeated oral care instruction to participants and staff (contact person) , supra gingival depuration if necessary. The group receive treatment each month.
  Interventions: Other: Intervention
- Control (No Intervention): Care as usual. Common oral hygiene help administered by nursing staff.

INTERVENTIONS:
Other: Intervention — Professional oral care
  Arms: Intervention

SUMMARY:
Today's increase of dentate elderly, many of them dependent, is a challenge, both according to the personal daily oral hygiene and dentistry. This is not only an oral problem, as research findings point to strong associations between oral and general health, even mortality. These findings are especially noticeable in elderly and frail individuals.

Dental care is usually performed in stationary dental clinics where the patients are transported to receive treatment. Dependent elderly dental patients may present many obstacles to traditional dental care due to cognitive limitations or dementia, mobility or transport problems. An alternative is domiciliary dental care where the dental staff performs the treatment by a home visit, in the patients daily living environment. The ability to handle personal oral hygiene is often decreased in these patients and left to overburdened nursing staff that often also lack sufficient knowledge about oral health care, why prophylactic professional oral care is especially important. This type of care can with rather simple equipments be performed as domiciliary treatment of good quality, while more advanced dental care may present restrictions in the home environment. However, in the Swedish dental system with subsidized dental care for dependent and elderly patients, there are restrictions for the number of prophylactic oral care treatments. The levels vary in different counties and regions. The rationale for this is probably tradition and economy as scientific evidence is lacking.

The aim with this project is to develop domiciliary professional oral care. The researchers will compare the effect of different regimens for domiciliary prophylactic professional oral care both according to content and frequency. The overall aim is to establish relevant recommendations for domiciliary prophylactic professional oral care.

DETAILED DESCRIPTION:
Background:

An increasing number of research publications point to the association between oral and general health. There are reports about associations between oral infections, coronary diseases, diabetes and respiratory tract infections but also between a high oral opportunistic micro flora and increased mortality in frail elderly individuals. It is important to develop oral care methods that effectively prevent the growth of an opportunistic micro flora and och oral diseases. Especially important is preventive methods in old and dependent individuals as these vulnerable patients groups have limited possibilities and access to relevant oral health care.

Professional oral care have been seen as an effective method to prevent dental diseases as caries and periodontal problems in elderly but in the new National guidelines for dentistry there is pointed to that there are no scientific proof for the effect of professional oral care, besides ordinary daily oral care in grownups. This conclusion could not be translated to frail elderly who are dependent on help from the nursing staff to receive or perform daily oral hygiene. The effect of domiciliary oral care have to our knowledge, not been explored. This type of care can with rather simple equipments be performed with good quality, while more advanced dental care may present more restrictions in the home environment. However, in the Swedish dental system with subsidized dental care for dependent and elderly patients, there are restrictions for the number of prophylactic oral care treatments. The levels vary in different counties and regions. The rationale for this is probably tradition and economy as scientific evidence is lacking.

Aim:

The aim is to develop and evaluate domiciliary prophylactic professional oral care. The researchers will compare the effect of different regimens for domiciliary prophylactic professional oral care on oral health in dependent elderly, both according to content and frequency. The overall aim is to to establish relevant recommendations for domiciliary prophylactic professional oral care.

Project plan:

Design:

The project is designed as a randomised, double blind, clinical study with two parallel study arms. Randomisation is performed at group level (ward unit), blind for the researchers and participants (allocation concealment). Data analysis will be made on individual level but presented at group level. Appliance for Ethical permission has been made and approved for the first part of the study that already is performed but it has to be completed with an approval for the continuing part of the study.

Pilot study:

Before the main clinical study started, a pilot study was performed in three months (half the time of the main study) to test the relevance of the study protocol, sample size but also the possible difference in oral health effects of hands-on-work including professional oral care compared to information and instruction. The pilot study was performed with 96 individuals included that randomly received professional oral care by a dental hygienist each month, information and re-instruction about oral care together with their daily care staff each month or served as a control. They all received baseline and effect registrations but with a selected number of variables that covered the purpose with the pilot study.

Participants The main study is planned to include 366 (2 x150 + 18 % compensation for estimated drop outs) dependent elderly individual in nursing homes. Inclusion criteria: at least 10 natural or fixed teeth inclusively osseointegrated implants, non smokers, ability to cooperate for oral assessment in 5-10 minutes and able to answer the Oral Health Related Quality of Life formula. Exclusion criteria: edentulousness and full dentures, cognitive limitations that is an obstacle for cooperation, malignancies and/or immunosuppressive diseases, coagulation defects. Anticoagulants will be registered but not as an exclusion criteria. The participants are consecutively recruited and sorted into the ward research group after informed consent - eventually with help of an advocate, (the ward research group is decided by chance when the first participant in the ward is recruited). A control group without any professional oral care during 6 months, will not be included in the main study, as it is not seen as good ethics to collect data without offer any oral care. Besides this, "ordinary care", either from the elderly themselves or nursing staff, vary. This is a confounding factor in the project that as far as possible is controlled by giving the same recommendations about routines for daily oral care to all included wards and participants. In accordance with ethical rules, the participants can interrupt their participation without explanation and negative consequences.

Sample size and power estimation:

The sample size is based on a power calculation of the least amount of individuals in each group to detect a significant difference of 7 % concerning bleeding at probing (BoP) between the groups (cluster randomisation in blocks on ward level to diminish unbalance in number of individuals in each ward), with risks for Type-I and Type-II estimated to alpha =0.05 and beta =0.20. For the primary effect variable, BoP (17), 150 individuals in each group are required. Due to high mortality in the study group (about 30 % in a year) and drop out because of illness, the sample will be increased with 18%. Accordingly, the number of participants will be n=366 (183 in each group). When drop outs, data analysis is performed due to intention-to-treat method.

Intervention:

All involved wards, nursing staff and relatives will be informed by a meeting where the project is presented and explained. At this occasion, a questionnaire will be distributed to the nursing staff to explore their knowledge and opinion about oral health care.

Standard rules for the daily oral hygiene during the study period will be set out. As far as possible, the oral care circumstances should be similar on each included study ward. Products containing chlorhexidine will be set out two weeks before the study start.

At baseline all participants will have an oral assessment together with a medical report including drug use, delivered by a registered nurse. On a subgroup consisting of 100 individuals (50 in each study arm), the oral micro flora is measured through sampling collected from supra gingival plaque with sterile toothpicks. The total number of microorganisms growing and the proportion of a) lactobacilli and streptococcus mutans and b) opportunistic bacteria including Staphylococcus aureus and candida are calculated.

As all participants is supposed to be eligible for free oral assessments at home and necessary dental care, their written oral care card will be updated with the routines that are actual during the study period. The exact performance of these routines will be established when the pilot study is evaluated.

Intervention in the research groups is professional oral care with electric tooth brush (Braun Oral-B), "ordinary" fluoridated tooth paste (1100-1450 ppm NaF), and repeated oral care instruction to participants and staff (contact person) supra gingival depuration if necessary, fluor varnish and delivery of saliva stimulating and replacing products to participants that show a stimulated salivation less than 1,0 ml/minute. All groups are continued during a period of 12 months. If electric tooth brush not is tolerated, an ordinary suitable tooth brush, chosen by the dental hygienist, will be used. Group A receive treatment each month, Group B receive no additional treatment (control).

Each participant is asked to brush their teeth every morning and evening with an "ordinary" fluoridated tooth paste (1100-1450 ppm NaF). Questions related to chewing ability and oral health related quality of life will be asked due to Geriatric Oral Health Assessment Index (GOHAI), as well as questions with the aim to evaluate how domiciliary professional oral care is experienced by the participants.

Clinical registrations due to study protocol (see below: effect variables), are performed by calibrated dental staff (dentists or dental hygienists) at baseline, after three months and after six months in all three study groups.

The dental staff will also have to get an opinion about the compliance of recommended routines and products with the help of questions to both the participants and the nursing staff. The exact construction of these questions will be made during the project period, as no validated formulas are available.

A coordinator will be required to monitor the including researchers concerning their commitment to the study protocol and to handle unforeseeable events, like patient safety, complaints, complications. Any treatment complications that are suspected or reported, will be registred and the project leader act upon a relevant way. If any participant is in need of dental care besides what the project activities can supply, this will also be reported to and handled by the project leader.

Effect variables:

Primary effect variable: bleeding on probing (BoP) in the gingival sulcus on buccal surfaces concerning the teeth 13, 12, 11, 21, 23, and 33, 32, 31, 41, 43 or the nearest comparable teeth. The bleeding will be scored at four levels (0-3) due to Modified Sulcus Bleeding Index. The measurements are performed at baseline and after three and each third month in both study groups. Comparison will be made on group level.

Secondary effect variables: Manifest caries is registred with the tooth as analysis unit DT Measurements are performed at baseline and each third month in both study groups.

Oral hygiene: Mucosal and plaque index, MPS, will be used both for fixed teeth and and partial removable dentures. The measurements are performed at baseline and each third month in both study groups..

Oral micro flora: The oral micro flora is measured through sampling collected from the same teeth as above mentioned according to BoP. The measurements are performed at baseline and each six month in both groups on the sub sample of 50 in each group.

Tertiary effect variables: Number of episodes with respiratory tract infections, pneumonia and use of antibiotics. Data is collected from a registered nurse. Measurements are performed at baseline and each six month in both groups.

Oral Health Related Quality of Life will also be measured by GOHAI, at baseline and each six month.

For the related nursing staff, two formulas will be used to measure knowledge about and attitudes to oral health, at baseline and each six month.

Significance:

Newly submitted data from professor Maude Wikström and her research group, inclusive main applicant Inger Wårdh, has pointed to that extensive oral hygiene routines may be effective in removing dental plaque but not opportunistic pathogens. This could probably be caused by oral dryness as the data also point to a need of stimulated flow at 1,0 ml/min before the pathogenic oral flora disappear, probably due to the self-cleaning effect of saliva. An important part of the professional oral health care would therefore be to supply with saliva stimulating or replacing products. Ongoing research also points to that we ought to use other products with the purpose to receive a higher pH-level in the oral cavity .It is lack of knowledge both according to content and frequency of professional oral care for dependent elderly and consequently neither how it ought to be subsidized from the government. However, in the first step it is important to create good routines for domiciliary professional oral care, which this project is able to do. The results will be published in scientific journals and also planned to be used in a PhD thesis and two master thesis.

ELIGIBILITY:
Inclusion Criteria:

* 10 or more natural teeth or fixed teeth inclusively osseointegrated implants
* non smokers,
* no or mild cognitive impairments

Exclusion criteria:

* severe cognitive impairments
* edentulousness and full dentures
* malignancies and/or immunosuppressive diseases, coagulation defects.

Anticoagulants will be registered but not as an exclusion criteria.

Ages: 80 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in bleeding on probing (BoP) each third month | 12 months
  Primary effect variable: bleeding on probing (BoP) in the gingival sulcus on buccal surfaces concerning the teeth 13, 12, 11, 21, 23, and 33, 32, 31, 41, 43 or the nearest comparable teeth. The bleeding will be scored at four levels (0-3) due to Modified Sulcus Bleeding Index. The measurements are performed at baseline and each third month up to 12 months in both study groups. Comparison will be made on group level.

SECONDARY OUTCOMES:
Changes from baseline in caries each third month | 12 months
  Manifest caries is registered with the tooth as analysis unit DT (decayed teeth). Measurements are performed each third month up to 12 months in both study groups.
Changes from baseline in Oral hygiene, each third month | 12 months
  Oral hygiene will be measured by Mucosal and plaque index. MPS, that will be used both for fixed teeth and and partial removable dentures. The measurements are performed at baseline and each third month up to 12 months in both study groups.
  The index is composed by a four level plaque score and a four level mucosal score that are added to a composed score in three levels: acceptable, unacceptable, bad
Changes from baseline in oral micro flora, each six month | 12 months
  Oral micro flora: The oral micro flora is measured through sampling collected from the same teeth as above mentioned according to BoP. The measurements are performed at baseline and each six month up to 12 months in both groups on the sub sample of 50 in each group.

OTHER OUTCOMES:
Changes from baseline in episodes with respiratory tract infections each six month | 12 months
  Number of episodes with respiratory tract infections, pneumonia and use of antibiotics. Data is collected from a registered nurse. Measurements are performed at baseline and each six month up to 12 months in both groups.
Changes from baseline in Oral Health Related Quality of Life, each six month | 12 month
  Oral Health Related Quality of Life will be measured by the validated index GOHAI, Geriatric Oral Health Assessment Index. Measurements are performed at baseline and each six month up to 12 months in both groups.
Changes from baseline in Knowledge within the nursing staff, each six months | 12 months
  The related nursing staff will be evaluated by a questionnaire that deals with the knowledge about oral health. Measurements are performed at baseline and each six month up to 12 months in both groups.
Changes from baseline in attitudes within the nursing staff, each six months | 12 months
  The related nursing staff will be evaluated by an index that deals with attitudes, the nursing DCBS (Dental Coping Beliefs Scale), to oral health. Measurements are performed at baseline and each six month up to 12 months in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Wårdh, Assoc prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinsk institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be be published in scientific papers but not on individual level, only group level